CLINICAL TRIAL: NCT01888523
Title: Stress Management for Cancer Survivors Using a Technologically Adapted Psychosocial Intervention: A Randomized Trial Determining the Effect of Expressive Writing on Psychoneuroimmunology Based Outcomes
Brief Title: Stress Management for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-14971
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Cancer Survivors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everyday experiences writing (Experimental): Involves logging in to an online survey and writing in the survey about your everyday experiences. This requires 20-30 minutes of writing a day for 4 consecutive days. You will also provide saliva samples.
  Interventions: Behavioral: Everyday experiences writing
- Expressive writing (Experimental): Involves logging in to an online survey and writing in the survey about your thoughts and feelings about your cancer. This requires 20-30 minutes of writing a day for 4 consecutive days. You will also provide saliva samples.
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Expressive writing — log in to an online survey and writing in the survey about your thoughts and feelings about your cancer. This requires 20-30 minutes of writing a day for 4 consecutive days. You will also provide saliva samples.
  Arms: Expressive writing
Behavioral: Everyday experiences writing — log in to an online survey and writing in the survey about your thoughts and feelings about your everyday experiences. This requires 20-30 minutes of writing a day for 4 consecutive days. You will also provide saliva samples.
  Arms: Everyday experiences writing

SUMMARY:
Determine the efficacy of a brief and inexpensive psychosocial intervention, (called expressive writing) in improving health outcomes for cancer survivors.

DETAILED DESCRIPTION:
This study aims to evaluate a computer-based stress-management therapy called expressive writing. This involves logging in to an online survey and writing in the survey about your thoughts and feelings about your cancer or to type in your everyday experiences. This requires 20-30 minutes of writing a day for 4 consecutive days. You will also provide saliva samples.

ELIGIBILITY:
Inclusion Criteria:

* have completed their cancer radiation treatment (intent to cure),
* are cancer free, i.e. do not have currently have a diagnosis of primary/secondary cancer or any recurrence/relapse of cancer,
* are in the re-entry phase of cancer survivorship, i.e. 2-12 months post-treatment completion,
* have access to a computer and internet in a private setting, e.g. at home,
* are fluent in English,
* are able to provide informed consent.

Exclusion Criteria:

* patients scheduled to undergo any type of cancer treatment (intent to cure/palliative) in the future (e.g. surgery after completing radiation),
* patients on any kind of corticosteroid medication (e.g. long-term prednisone therapy),
* patients having any condition that affects function of the adrenal glands (e.g. adrenal hyperplasia),
* patients with limited ability to produce saliva, e.g. patients that received radiation (or surgery) on the face region or on salivary glands; or patient's suffering from dry mouth (e.g. Sjögren's syndrome),
* patient's suffering from inflammation of the oral cavity (e.g. gingivitis).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
salivary cortisol levels | Up to 6 weeks
  Participants will be asked to give their saliva samples through chewable swabs 3 times per day on every day of data collection, i.e. once at baseline, which is 24 hours before the intervention, and twice after the intervention, specifically, 24 hours and 6 weeks post-intervention. Participants will be requested to chew on their swabs and spit into their containers at the following times: 1) immediately after waking up, 2) within 30 min after waking, and 3) immediately before going to sleep.

SECONDARY OUTCOMES:
salivary α-amylase and C-Reactive Protein (CRP) | Up to 6 weeks
  Participants will be asked to give their saliva samples through chewable swabs 3 times per day on every day of data collection, i.e. once at baseline, which is 24 hours before the intervention, and twice after the intervention, specifically, 24 hours and 6 weeks post-intervention. Participants will be requested to chew on their swabs and spit into their containers at the following times: 1) immediately after waking up, 2) within 30 min after waking, and 3) immediately before going to sleep.
self-reported psychometric measures | Up to 6 weeks
  The levels of perceived psychological stress levels will be assessed using the Perceived Stress Scale (PSS). This psychometric instrument has 14 items (see Appendices) that will be answered by the participants on a 5-point Likert scale. This scale has a demonstrated good reliability in healthy and clinical populations, and has a Chronbach's alpha value of 0.86109.
  The severity of fear of cancer recurrence (FCR) is a good indicator for the level of negative emotional stress experienced. FCR Instrument is a 42 item multi-dimensional measure which specifically describes the amount of emotional stress experienced.
  Cancer Behavior Inventory-Brief Version (CBI-B), a 12 item self-reported instrument to measures the level of self-efficacy among Cancer Survivors for their capacity to cope with cancer. All 12 items are rated on a 9-point likert scale that ranges from 1 ("not all confident") to 9 ("totally confident").

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brown, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States